CLINICAL TRIAL: NCT07270003
Title: A Prospective, Single-arm, Open-label Clinical Trial to Evaluate the Efficacy and Safety of Ivarmacitinib in the Treatment of Palmoplantar Pustulosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20252406-C-1
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-09

CONDITIONS: Palmoplantar Pustulosis (PPP)
MeSH Terms: conditions — Psoriasis | interventions — ivarmacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral ivarmacitinib 4mg once daily for 12 weeks (Other)
  Interventions: Drug: Ivarmacitinib

INTERVENTIONS:
Drug: Ivarmacitinib — Oral ivarmacitinib 4mg once daily for 12 weeks

SUMMARY:
What's the problem? Palmoplantar pustulosis (PPP) is a long-term skin condition that mainly affects the palms of hands and soles of feet. It causes red, scaly skin with small, non-infectious blisters (called pustules), and often brings pain, itching, or even joint damage over time. It's more common in women aged 40-58 and makes daily life harder. Right now, treatments for PPP aren't great. Creams (like corticosteroids) make symptoms come back fast. Pills (such as acitretin) work slowly, don't always help, and can have bad side effects. Some strong injectable drugs (biologics) are expensive, need long-term use, and require regular checks for infections-plus they don't work well for many PPP patients.

What's this study trying to do?

This study will test a new pill called ivarmacitinib to see if it works for PPP, and if it's safe. Here's what researchers want to find out:

Does ivarmacitinib reduce PPP symptoms (like blisters and redness)-and how quickly? Does it help with joint problems that sometimes come with PPP? Are there side effects (like infections, headaches, or stomach issues)? And how common or serious are they? Do things like a patient's age, past treatments, or other health issues affect how well ivarmacitinib works? How will the study work? This is a open study (everyone knows they're taking ivarmacitinib) with 60 patients at the First Affiliated Hospital of Air Force Medical University (China).

Who can join? Must be 18 or older, with a confirmed PPP diagnosis. Tried at least one other standard treatment (like pills or creams) that didn't work or caused too many side effects.

Must not have serious health issues like active infections (e.g., tuberculosis, hepatitis), low blood cell counts, or bad liver/kidney problems.

What will patients do? Take one 4mg ivarmacitinib pill every day for 12 weeks. Can't use other drugs or light therapy for PPP during this time (but simple moisturizers or meds for other health issues are okay).

Before the study starts: Doctors will check basic health (age, weight, lifestyle), PPP symptoms, and do blood tests, urine tests, and a chest X-ray.

During the study (Weeks 1, 2, 4, 8, 12): Doctors will check how symptoms are changing, ask if patients have any side effects, and do another round of blood tests at Week 12.

What will researchers look for? Does it work? The main goal is to see how many patients have a 50% or bigger reduction in PPP symptoms by Week 12. They'll also check if symptoms get 75% or 90% better, if joints feel better, and if daily life (like working or sleeping) improves.

Is it safe? Researchers will track all side effects-especially infections, blood clots, stomach aches, or headaches-and how serious they are.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old; clinically/pathologically confirmed PPP; failure/intolerance to ≥1 conventional systemic therapy (12-24 weeks of standard dosing); physician-judged suitability for ivarmacitinib; signed informed consent.

Exclusion Criteria:

* Lymphocyte count <0.5×10⁹/L, neutrophils <1×10⁹/L, platelets <100×10⁹/L, or hemoglobin <80g/L; serum creatinine >132.6μmol/L, AST/ALT >2×ULN, or total bilirubin >2.0mg/dL; active infections (tuberculosis, hepatitis B/C, systemic candidiasis); other conditions hindering participation or data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
PPPASI50 response rate (≥50% reduction in PPPASI score) | Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided